CLINICAL TRIAL: NCT01389674
Title: Hybrid Intraprocedural Imaging From 2D-Strain-echocardiography and X-ray Based Biplane Coronary Angiography for Guiding Interventional Revascularization Therapy
Brief Title: Hybrid Intraprocedural Imaging Based on 2 Different Imaging Methods
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HIB-Study; CTC-A 08-001; EK 079/10
Record Dates: First submitted 2009-02-03; First posted 2011-07-08 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Angina Pectoris; Left Ventricular Wall Motion Abnormalities
Keywords: coronary stenosis; Angina pectoris; left ventricular wall motion abnormalities
MeSH Terms: conditions — Angina Pectoris; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2D-strain echo (Experimental): After myocard vitality diagnostics with MRI follows a stress echocardiography to determine the LV volumes and EF. The received Data are compare with the MRI-Data(reference)to identify the ideal strain-parameters and Cut-Off-Result for an intraprocedural vitality diagnostic of the different films (endocardial, myocardial and epicardial).
  Interventions: Procedure: 2D-strain echo

INTERVENTIONS:
Procedure: 2D-strain echo — 2D-strain-analysis with elevation of the radial and circumferential strain and strain rate parameter(systolic and diastolic)occurs through the echocardiography.
  Comparison of the echocardiography and the MRI-vitality data, calculation of a cut out of vision value of a vitality diagnosis with the help of 2D-strain-analysis.

SUMMARY:
The investigators will check the feasibility of an intraprocedural vitality diagnostics and the identification of an indication for Percutaneous transluminal coronary angioplasty (PTCA).

DETAILED DESCRIPTION:
After myocard vitality diagnostics with MRI patients will underwent additionally an stress echocardiography within the exploration. By this ultrasound we will measure the LV mass and the ejection fraction per apical 2-, 3- and 4-chamber view.

In addition a 2D-strain-analysis will be done to measure the systolic and diastolic strain and also the circumferential and radial strain rate parameter (by depicting three parasternal short axis views in the basal, mid-ventricular and apical plane).

These measurements will be compared with the studies-conditioned MRI-finding (as reference) to find the optimal strain-parameter and the optimal cut-off-data for an intraprocedural vitality diagnostics of the single layers (endocardial, myocardial, and epicardial) for this patient group.

The data upraised through this are compared off-line to the MRI findings.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular wall motion abnormalities
* existent myocardial vitality MRI exploration
* reduced LV-function
* steady angina pectoris
* patients which are legally competent and which are mentally able to understand the study staff
* patients give their written consent

Exclusion Criteria:

* pregnancy or lactation
* acute or instable angina pectoris
* acute myocardial infraction in the last 3 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cut-Off-Value of vital myocardial tissue | time during hospitalization
  It will be determine cutt-off-value of vital myocardial tissue in comparison to MRI myocardial vitality findings.

SECONDARY OUTCOMES:
feasibility and safety of echocardiography during catheter investigations | time during hospitalization and 1 months afterwards
  it will be analyzed if it is logistically possible to perform echo-test during the actual catheter investigations (feasibility) and if the patient will be exposed to any safety risk for logistic or sterility reasons.
Determination of Strain-Parameter for identification of vital myocardial tissue | time during hospitalization
  It will be determitated optimal Strain-Parameter(circumferential, systolic or diastolic)for identification of vital myocardial tissue

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, MD, Principal Investigator — RWTH Aachen University
Locations (1):
- University Hospital Aachen, Aachen, Germany